CLINICAL TRIAL: NCT00715065
Title: Neuroimaging in Blood Phobia Syncope
Brief Title: fMRI in Blood Phobia Syncope
Status: Withdrawn | Type: Observational
Why Stopped: Could not get funding for fMRI studies at this time.
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Satish R. Raj, Assistant Professor, Vanderbilt University
Other Study IDs: 080608; NIH UL1 RR024975
Record Dates: First submitted 2008-07-10; First posted 2008-07-15 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Syncope; Blood Injury Phobia; Autonomic Dysfunction
Keywords: syncope; faint; blood; blood injury phobia; phobia
MeSH Terms: conditions — Syncope; Primary Dysautonomias; Phobic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: Healthy control subjects (who do not faint at the sight of blood)
  Interventions: Procedure: fMRI Scan
- 1: People who faint at sight of blood
  Interventions: Procedure: fMRI Scan

INTERVENTIONS:
Procedure: fMRI Scan — Subjects will undergo a functional MRI scan of the head lasting ~45 minutes. They will be repeatedly shown video clips of blood, other disgusting things, or are neutral.

SUMMARY:
We plan to study patient who faint in response to the sight of blood and compare them to healthy subjects who do not. We are going to use a special type of MRI scan (functional MRI) to determine if there are differences in brain activation in response to seeing bloody or gory pictures that occur before the fainting occurs.

DETAILED DESCRIPTION:
Another aim of the study is to determine whether or not differences in personality traits among people with blood phobia is associated with differences in BOLD signal responses during fMRI.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* 1. History of at least one syncopal episode upon exposure to viewing blood (Case Group)
* Negative urine pregnancy test on study day

Exclusion Criteria:

* Vasoactive medications (within 2 weeks of study day)
* antihypertensives
* beta blockers
* vasoconstrictors
* Psychotropic medications (within 4 weeks of study day)
* History of psychostimulant or opiate use
* History of alcohol, benzodiazepine or cannabis abuse or dependence

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Patients with at least 1 prior syncopal episode in response to viewing blood
  2. Healthy subjects without a history of syncope
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
fMRI BOLD signal | Immediate

SECONDARY OUTCOMES:
Blood Injection Symptoms Scale | Single visit
Disgust Scale (Revised) | Single Visit

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Autonomic Dysfunction Center, Nashville, Tennessee, United States